CLINICAL TRIAL: NCT00005920
Title: A Multiclinic, Double-Blind, Randomized, Dose-Comparison Study to Evaluate the Safety, Tolerability, and Efficacy of L-743,872 in the Treatment of Fluconazole-Unresponsive Oropharyngeal Candidiasis in Adults
Brief Title: Safety and Effectiveness of Giving L-743,872 to Patients With Thrush That Has Not Been Cured With Fluconazole
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 267B; 012-00
Record Dates: First submitted 2000-06-19; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-06

CONDITIONS: Candidiasis, Oral; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Dose-Response Relationship, Drug; Fluconazole; Antifungal Agents; Candidiasis, Oral; Pharyngeal Diseases; MK 0991
MeSH Terms: conditions — Candidiasis, Oral; HIV Infections; AIDS-Related Opportunistic Infections; Pharyngeal Diseases | interventions — Caspofungin

INTERVENTIONS:
Drug: L-743,872

SUMMARY:
The purpose of this study is to see if it is safe and effective to give L-743,872 to patients with thrush, an AIDS-related yeast infection of the mouth, that has not been cured with fluconazole treatment.

DETAILED DESCRIPTION:
Patients are randomized to treatment with L-743,872 at one of two doses administered intravenously by a peripheral line once-daily. Patients are treated for 48 hours beyond resolution of symptoms or for a maximum of 14 days. Each patient is expected to complete the study, including the 14-day follow-up, within approximately 4 weeks. A physical examination is performed daily during the antifungal treatment period and at the follow-up visits 7 and 14 days post-therapy. Laboratory tests of blood and urine for safety are performed every three days during treatment and at follow-up 7 days post-therapy. Liver enzymes are drawn at the 14-day follow-up visit.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Have thrush that has not responded to fluconazole treatment.
* Are 18-65 years old.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70

CONTACTS AND LOCATIONS:
Locations (1):
- Carol Sable, Rahway, New Jersey, United States